CLINICAL TRIAL: NCT06391554
Title: Effects of EDUcation and EXercise Compared to Education Alone on Clinical and Physiological Outcomes in Patients With Hip Osteoarthritis
Acronym: EDUEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Silkeborg (Other); Vejle Hospital (Other); Physiotherapy Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EDUEX
Record Dates: First submitted 2024-04-22; First posted 2024-04-30 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRT + EDU (Experimental)
  Interventions: Other: PRT; Other: EDU
- EDU (Active Comparator)
  Interventions: Other: EDU

INTERVENTIONS:
Other: PRT — An initial 12-week exercise intervention, consisting of 1-hour group sessions of progressive resistance training supervised by a physiotherapist 2 times per week. The sessions consist of a 10-minute submaximal warm up on an exercise bike followed by 50 minutes of PRT with exercises targeting the muscles of the hip and knee joints; leg press, hip extension, hip abduction, hip flexion and knee extension. The progression will be in line with guidelines provided by the American College of Sports Medicine. The intensity will follow repetition maximum (RM) targets, from 12 RM for the first week towards 8 RM for the last weeks. After the 12 weeks, participants will receive 8 booster sessions and are given a membership to a fitness center where they will be encouraged to continue the exercise program on their own.
  Arms: PRT + EDU
Other: EDU — Three EDU sessions provided by a trained physiotherapist involving important disease-specific information. The sessions will address knowledge of OA, treatment options with a specific focus on physical activity recommendations, advice on self-management and more. All three sessions will emphasize on engaging the participants actively and sharing experiences with each other.

SUMMARY:
The EDUEX trial will determine whether the addition of progressive resistance training (PRT) to a patient education program (EDU) will improve clinical outcomes in patients with hip OA.

In a subsample, the effect of PRT on the articular cartilage and other structures of the hip joint is investigated. In this subsample, a comprehensive assessment of possible mechanisms underlying the effects of exercise on pain and function is undertaken.

The EduEx trial will be a multicentre, stratified (by site), block randomized (allocation 1:1), controlled, parallel-group superiority trial. 150 people with hip OA will be recruited from hospitals, physiotherapy clinics, social media and newspapers. Participants will be randomized to PRT and EDU or EDU alone. All 150 participants will be included in the clinical evaluation study (CLIN). The last 40 participants randomized to PRT+EDU and to EDU, respectively, will also be included in the mechanistic (MECH) evaluation study (n=80), by being asked to participate in additional outcome assessments. The primary endpoint will be the 12 months follow-up for both the CLIN and MECH study, while a secondary endpoint will be the 3-month follow-up.

DETAILED DESCRIPTION:
DESIGN

The EduEx trial will be a multicentre, stratified (by site), block randomized (allocation 1:1), controlled, parallel-group superiority trial. 150 people with hip OA will be recruited from the Orthopedic Departments at hospitals and from physiotherapy clinics, social media and newspapers. Participants will be randomized to PRT+EDU or EDU.

All 150 participants will be included in the clinical evaluation study (CLIN) while only the last 40 participants randomized to PRT+EDU and EDU, respectively, will also be included in the mechanistic evaluation study (MECH, n=80), by being asked to participate in additional outcome assessments including magnetic resonance imaging of the hip.

The primary endpoint will be the 12 months follow-up for both the CLIN and MECH study, while the secondary endpoint will be the 3-month follow-up.

RANDOMIZATION

After baseline assessment, participants will be randomized in a 1:1 ratio to PRT+EDU or EDU. A computer-generated list of random numbers will be generated in the Research Electronic Data Capture (REDCap) system. The randomization will be stratified by site and block randomized, to ensure equal distribution of allocations among trial sites. Two lists of random numbers will be generated, one for the first 70 participants and one for the last 80 participants recruited, to enable an even distribution of treatment allocation of the 80 participants in the MECH subsample. Treatment allocation will be concealed as one of the principal investigators will use the randomization tool only after the baseline assessment has been performed.

INTERVENTIONS

The PRT and EDU interventions will be conducted either at the collaborating hospital departments or physiotherapy clinics across Denmark.

PRT: Participants allocated to receive PRT will attend 3 months of supervised PRT followed by 9 months of unsupervised PRT with the addition of 8 exercise booster sessions. The PRT program consists of two weekly training sessions (60 min per session) with ≥48 hours of rest between sessions. All supervised PRT sessions will be group-based (up to 5 participants) supervised by one physiotherapist.

EDU: Both treatment arms will attend three EDU sessions provided by a trained physiotherapist involving important disease-specific information. The sessions will address knowledge of OA, treatment options with a specific focus on physical activity recommendations, advice on self-management and more. All three sessions will emphasize on engaging the participants actively and sharing experiences with each other.

STATISTICAL ANALYSIS PLAN

The analyses will be based on the between-group difference in change in the primary and secondary outcomes from baseline to the 12 months follow-up, according to the intention-to-treat (ITT) principle. Additionally, per protocol analyses will be performed including only participants with high adherence to the EDU sessions (at least 2 sessions attended) and high adherence to the exercise sessions (≥80% of the planned sessions completed) and high exercise fidelity (≥80% of prescribed repetitions performed). Between-group comparisons of change from baseline to follow-up in the primary and secondary continuous outcomes will be analysed using a repeated measures mixed model with participants and sites as random effects and with visits and treatment arm as fixed effects.

DATA MANAGEMENT

All data and outcomes collected from participants will be entered into the REDCap database. For the patient reported outcomes, participants will fill out questionnaires directly into REDCap. If a participant is unable to do so, they will fill out paper versions of the questionnaires and the tester will enter it into REDCap and shred the paper versions. The data will be maintained in storage for five years after trial termination.

PATIENT AND PUBLIC INVOLVEMENT

In the EduEx trial we have established an advisory board of four patients with hip osteoarthritis and a physiotherapists. Patients and physiotherapists have been invited to participate in the board throughout the research project. The board have and will continue to influence clinical outcomes, practicalities, and content of the interventions. The board will have one meeting every three months during the planning, conducting and dissemination processes of the trial and will give advice (consultation level of involvement) throughout.

ETHICAL CONSIDERATIONS

The study intervention is non-invasive and is expected to result in a generally optimized health status of the included participants. Approval from the Central Denmark Region Committee on Health Research has been obtained for the EduEx trial. Written informed consent will be obtained from all participants prior to inclusion and the project will be performed in accordance with the Helsinki Declaration. Authorship eligibility will be based on the recommendations from The International Committee of Medical Journal Editors. Any important protocol amendments for The EduEx trial will be registered at ClinicalTrial.gov and reported to the Central Denmark Region Committee on Health Research.

RESEARCH RESULTS

The results from this trial will be published in peer-reviewed scientific journals and presented at congresses, regardless of whether the results are inconclusive, negative or positive.

There are 3 preplanned studies to be conducted on the results from this trial that will be reported in 3 separate research papers:

1. The primary clinical evaluation study (CLIN) comparing effects of PRT+EDU and EDU alone on the primary outcome of HOOS ADL is study number one.
2. The primary mechanistic evaluation study (MECH) comparing PRT+EDU and EDU alone on changes in hip joint tissue is study number two.
3. A secondary MECH evaluation study (MECH2) is study number three, in which the mechanisms of exercise are investigated by looking at associations of changes in other outcomes with the changes seen for hip pain and physical function.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with hip OA according to the criteria by the National Institute for Health and Care Excellence (NICE)
* Radiographic verification of hip OA diagnosis with Kellgren Lawrence score of 2 or 3 in one or both hips
* Not scheduled for a total hip replacement within the following 12 months
* An event of hip pain every day of at least 3 out of 10 on a numerical rating scale during the last 14 days
* Age ≥ 45 years
* Adequacy in written and spoken Danish

Exclusion Criteria:

* Comorbidity that markedly influences hip function or degeneration of tissue in or around the hip joint (rheumatic, neurological, mental or other)
* Surgery in the lower extremities within the six months prior to inclusion
* BMI > 40
* Pregnancy
* Resistance exercise (weights or elastic bands) for the lower extremities exceeding 12 sessions over the last 6 months or 6 sessions over the last 3 months
* Suffering from claustrophobia or not tolerating whole body MRI scanner
* Metallic implants from the waist to just above the knee
* Pacemaker or other medical devices that are not MR approved

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline to 12 month follow-up (primary endpoint) in the Hip Disability and Osteoarthritis Outcome Score (HOOS) ADL function subscale | Measured at baseline, 12 weeks and 12 month follow-up
  Primary outcome for the CLIN study and secondary outcome for the MECH study. The HOOS ADL function subscale is a 17-item patient-reported outcome measure designed to assess ADL function in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better ADL function status.
Changes from baseline to 12-month follow-up (primary endpoint) in the hip articular cartilage of the index hip measured by MRI T2 relaxation time mapping. | Measured at baseline and 12 month follow-up
  Primary outcome for the MECH study

SECONDARY OUTCOMES:
Changes in the Scoring Hip Osteoarthritis with MRI (SHOMRI) semiquantitative scoring system for evaluating imaging features relevant to the severity and progression of osteoarthritis | Measured at baseline and 12 month follow-up
  Key secondary outcome for the MECH study. The scoring system cardinal features related to osteoarthritis of the hip joint on a scale of 0-5 (where 5 is most severe). These features are: articular cartilage loss, bone marrow edema pattern, subchondral cysts, labral abnormality, paralabral cysts, intra-articular bodies, effusion/synovitis and ligamentum teres abnormality.
Change in the HOOS Pain subscale | Measured at baseline, 12 weeks and 12 month follow-up
  Key secondary outcome for the CLIN study and for the MECH study. The HOOS pain subscale is a 10-item patient-reported outcome measure designed to assess hip pain in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better pain status.
Change in the HOOS Hip-related Quality of Life subscale | Measured at baseline, 12 weeks and 12 month follow-up
  Key secondary outcome for the CLIN study and secondary outcome for MECH study. The HOOS quality-of-life subscale is a four-item patient-reported outcome measure designed to assess hip-related quality-of-life in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better quality-of-life status.
Changes from baseline to 12-month follow-up (primary endpoint) in the articular cartilage of the index hip measured by MRI T1rho relaxation time mapping. | Measured at baseline and 12 month follow-up
  Secondary outcome for the MECH study.
  This outcome was changed from co-primary to secondary outcome on 09/17/2025 where 68 participants had been included in the trial and no MECH participant was included or had attended baseline assessment. As such, no MRI scans had been conducted for trial participants at this time. This change was made due to persistent technical issues with the T1r MRI scanning sequence resulting in a high risk of missing data for this outcome.
Change in the HOOS Symptoms subscale | Measured at baseline, 12 weeks and 12 month follow-up
  Secondary outcome for the CLIN study and MECH study. The HOOS symptoms subscale is a five-item patient-reported outcome measure designed to assess other hip symptoms in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better symptoms status.
Change in the HOOS Sport/recreation subscale | Measured at baseline, 12 weeks and 12 month follow-up
  Secondary outcome for the CLIN study and MECH study. The HOOS sports and recreation subscale is a four-item patient-reported outcome measure designed to assess sports and recreation function in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better sports and recreation status.
Change in the 30 second chair stand test | Measured at baseline, 12 weeks, and 12 month follow-up
  Secondary outcome for the CLIN study and exploratory outcome for MECH study. The 30s-CST is a physical function test designed to assess sit-to-stand function (number of repetitions).
Change in the 9-step stair climb test | Measured at baseline, 12 weeks, and 12 month follow-up
  Secondary outcome for the CLIN study and exploratory outcome for MECH study. Measures time (in seconds) taken to negotiate 9 steps on a standard step-height stair-way (up and down).
Change in the 40 meter fast-paced walk test | Measured at baseline, 12 weeks, and 12 month follow-up
  Secondary outcome for the CLIN study and exploratory outcome for MECH study. The 40m-FPWT is a physical function test designed to assess short distance maximum walking speed.
Number of treatment responders according to OMERACT-OARSI response criteria | Measured at 12 weeks and 12 month follow-up
  Secondary outcome for the CLIN study. The criteria are:
  1. In either pain (HOOS pain subscale) or function (HOOS ADL function subscale), a high improvement in the subscale, where high improvement in a subscale is achieved if there is both a > 50% improvement from Baseline and an absolute change from Baseline of > 20 points (0-100 scale), OR
  Improvement in at least two of the following three:
  Improvement in pain (HOOS pain subscale) defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 points (0-100 scale) Improvement in function (HOOS ADL function subscale) defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 points (0-100 scale) Improvement in patient's global assessment defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 mm (0-100 scale)

OTHER OUTCOMES:
Demographic data consisting of sex, age, weight, height, BMI, analgesics, cohabiting status, marital status, employment status, alcohol intake, smoking habits, duration and severity of symptoms, current and previous treatment, co-morbidities. | Measured at baseline (treatment received, weight, co-morbidities, and analgesic use is also measured at 12 weeks and 12 month follow-up
  Descriptive data for CLIN study and MECH study
Safety outcomes will include number of adverse events and serious adverse events (SAE) | Recorded throughout the trial (up to 1 year)
  Descriptive data for CLIN study and MECH study. SAE are defined according to the International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) guidelines.
Participants who drop out from the trial | Recorded throughout the trial (up to 1 year)
  Descriptive data for CLIN study and MECH study
Adherence to PRT exercise program | Recorded throughout the trial (up to 1 year)
  Descriptive data for CLIN study and MECH study. Recorded as attendance to each session (yes/no) and presented as number of and proportion of sessions attended
Adherence to EDU sessions | Recorded throughout the trial (up to 1 year)
  Descriptive data for CLIN study and MECH study. Recorded as attendance to each session (yes/no) and presented as number of and proportion of sessions attended
Fidelity to the PRT exercise program | Recorded throughout the trial (up to 1 year)
  Descriptive data for CLIN study and MECH study. Recorded as number of exercise repetitions and sets completed and presented as numbers and proportions
Patient expectations for treatment modalities | Measured at baseline
  Exploratory outcome for the CLIN study and MECH study. Participants are asked to rate their expected benefit from the study interventions on a questionnaire with a 5 point scale (very little or no improvement to very large or complete improvement).
Patient preferred treatment option | Measured at baseline
  Exploratory outcome for the CLIN study and MECH study. Participants are asked to list the treatment options they would prefer on a questionnaire with 10 options and the additional option of adding a free text description of a treatment not pre-specified.
Change in the Pain Catastrophizing Scale | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study. Participants rate their agreement with 13 statements on a scale from 0 to 4 (0=not at all, 4=to a very large extent).
Change in the Hospital Anxiety and Depression Scale | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study
Number of painful sites on a region-divided body chart | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study
Change in dietary pattern measured by the danish "Hjertekost" questionnaire | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study. Dietary intake is rated in two categories "fat" and "fish, greens and fruit" on a scale from 0-100 (higher score indicates better dietary pattern)
Patient-reported Global Perceived Effect | Measured at 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study. Perceived effect of interventions is rated on a 7 point likert scale from significantly worse to significantly better.
Patient-reported Treatment Failure of the interventions | Measured at 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study. Participants are asked if they think the treatment has failed (yes/no).
Change in the Self-Efficacy for Managing Chronic Disease 6-item Scale | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study. Participants are asked to rate their self-perceived self-efficacy from a scale from 1 to 10 (higher score means better outcome) by a 6 item questionnaire
Change in the Pittsburgh Sleep Quality Index | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study. The questionnaire rates the sleep quality on a global score ranging 0 to 21 (higher scores indicate worse sleep quality)
Changes in physical activity level measured by accelerometry | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study. The number of minutes spent each day in sedentary, moderate intensity and vigorous intensity activity is measured.
Treatment response according to the Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) criteria | Measured at 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study. Each participant is rated as a responder or non-responder in respect to the OMERACT-OARSI criteria.
Changes in pain sensitivity using quantitative sensory testing by a computer-controlled cuff algometer. | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study
Changes in pain tolerance thresholds using quantitative sensory testing by a computer-controlled cuff algometer. | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study
Changes in temporal summation using quantitative sensory testing by a computer-controlled cuff algometer. | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study
Changes in conditioned pain modulation using quantitative sensory testing by a computer-controlled cuff algometer. | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study
Changes in maximal voluntary isometric contraction by Isokinetic dynamometry. Assessed for hip flexors and extensors, and knee flexors and extensors. | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study
Changes in rate of force development by Isokinetic dynamometry. Assessed for hip flexors and extensors, and knee flexors and extensors. | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study
Changes in maximal voluntary muscle activation using the interpolation twitch technique. | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the MECH study
Changes in anatomical cross-sectional area of m. Quadriceps, Gluteus Maximus and Gluteus Medius measured by MRI cross-sectional area | Measured at baseline and 12 month follow-up
  Exploratory outcome for the MECH study
Changes in extramyocellular infiltrations of fat and connective tissue of m. Quadriceps, Gluteus Maximus and Gluteus Medius measured by MRI cross-sectional area | Measured at baseline and 12 month follow-up
  Exploratory outcome for the MECH study
Changes in bone mineral density measured by Dual energy xray absorptiometry | Measured at baseline and 12 month follow-up
  Exploratory outcome for the MECH study
Changes in muscle mass measured by Dual energy xray absorptiometry | Measured at baseline and 12 month follow-up
  Exploratory outcome for the MECH study
Changes in fat mass measured by Dual energy xray absorptiometry | Measured at baseline and 12 month follow-up
  Exploratory outcome for the MECH study
Changes in concentrations of blood serum biomarkers for low grade systemic inflammation, cartilage degradation, cartilage formation, bone degradation, and synovial inflammation. | Measured at baseline and 12 month follow-up
  Exploratory outcome for the MECH study. The blood serum concentration of the following biomarkers will be assessed: C-RP, CTX-II, PRO-C2, C1M, MMP-3, PIIANP, sCOMP, and sHA
Changes in hip pain assessed by a numerical rating scale from 0-10 (0 = no pain, 10 = worst imaginable pain) | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study
Changes in One-legged 30 second chair stand test measured for index leg and contralateral leg | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study
Changes in indirectly measured VO2max by the Åstrands submaximal cycle test | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study
Changes in patients global assessment of impact of osteoarthritis | Measured at baseline, 12 weeks, and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study. Impact is assessed by a 0-100 mm visual analog scale (higher score means worse outcome)
Patient Acceptable Symptom State (PASS) | Measured at 12 weeks and 12 month follow-up
  Exploratory outcome for the CLIN study and MECH study. Participants are asked on a questionnaire whether they think their current symptom state is satisfactory (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Troels Kjeldsen, MSc, Principal Investigator — Aarhus University Hospital; Thomas Frydendal, PhD, Principal Investigator — Aarhus University Hospital; Inger Mechlenburg, Prof., Study Director — Aarhus University Hospital; Ulrik Dalgas, Prof., Study Director — University of Aarhus
Locations (2):
- Denmark (2):
  - Aarhus University, Aarhus C
  - Aarhus University Hospital, Aarhus N

IPD SHARING:
Plan to Share IPD: Yes
Anonymised patient-level data will be made available if required by the scientific journal, in which the results of the trial are published. Additionally, researchers presenting a justified cause for receiving the data can obtain it after a data access agreement has been signed.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after publication of the trial
Access Criteria: Data access will be reviewed by the author group. Requesters will be required to sign a data access agreement.